CLINICAL TRIAL: NCT06221761
Title: A Prospective Randomized Controlled Study on the Prophylactic Use of Antibiotics Within 72 Hours After Acute Burn Injury in Patients
Brief Title: A Study on the Prophylactic Use of Antibiotics Within 72 Hours After Acute Burn Injury in Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20231226
Record Dates: First submitted 2023-12-26; First posted 2024-01-24 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2023-12

CONDITIONS: Burn Infection
Keywords: burn; infection; antibiotic
MeSH Terms: conditions — Burns; Infections

STUDY DESIGN:
Intervention Model Description: Participants will be randomly divided into two groups, one using antibiotics and the other not using antibiotics
Who Masked: Participant
Masking Description: Participants do not know which group they will be assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non antibiotic group (Experimental): Not using antibiotics within 72 hours after burns
  Interventions: Drug: not using antibiotic
- antibiotic group (Active Comparator): Using antibiotics within 72 hours after burns
  Interventions: Drug: using antibiotic

INTERVENTIONS:
Drug: not using antibiotic — no antibiotic application
  Arms: Non antibiotic group
Drug: using antibiotic — antibiotic application
  Arms: antibiotic group

SUMMARY:
The goal of this clinical trial is to compare in acute burn patients.

The main question it aims to answer are:

• what is the impact of early prophylactic use of antibiotics on prognosis Participants will be randomly divided into an antibiotic group and a non antibiotic group.

Researchers will compare the two groups to see the 72 hour wound bacterial culture negative rate.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form
* Promise to comply with research procedures and cooperate with the implementation of full process research
* Age 18 and above
* Emergency hospitalization of patients in the burn department, within 24 hours after injury
* No immunodeficiency disease, no history of using immunosuppressive drugs, no antibiotics being used or infectious diseases at the time of admission
* If a woman is in the reproductive period, she should not be pregnant

Exclusion Criteria:

* Unable to obtain informed consent from subjects, family members, or authorized agents
* At the time of admission, antibiotics were being administered
* During pregnancy
* Presence of infectious diseases before admission
* Existence of immunodeficiency diseases or use of immunosuppressive drugs
* The subjects are currently undergoing other clinical studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Negative rate of bacterial culture | hour 72
  Number of cases with negative wound culture bacteria/total number of cases

SECONDARY OUTCOMES:
28 day mortality rate | 28 day after burn
  28 day mortality rate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] ISBI Practice Guidelines Committee; Steering Subcommittee; Advisory Subcommittee. ISBI Practice Guidelines for Burn Care. Burns. 2016 Aug;42(5):953-1021. doi: 10.1016/j.burns.2016.05.013. PMID 27542292
- [Result] Avni T, Levcovich A, Ad-El DD, Leibovici L, Paul M. Prophylactic antibiotics for burns patients: systematic review and meta-analysis. BMJ. 2010 Feb 15;340:c241. doi: 10.1136/bmj.c241. PMID 20156911